CLINICAL TRIAL: NCT04299763
Title: Oat β-glucans as a Supplement in Chilean Subjects With Type 2 Diabetes for Metabolic Control
Brief Title: Oat Beta-glucan as a Supplement in Chilean Type 2 Diabetics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro de Estudios en Alimentación y Nutrición, Chile (Other)
Responsible Party: Principal Investigator, José Luis Pino Villalón, Nutritionist, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DOCNUTAL
Record Dates: First submitted 2019-09-17; First posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Type2 Diabetes
Keywords: beta-Glucans; Diabetes Mellitus, Type 2; Chile
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — beta-glucan, (1-3)(1-4)-

STUDY DESIGN:
Intervention Model Description: Two groups were used: experimental (n 17): they received oat beta-glucan supplement to be added to breakfast (5 g). Control group: they received a placebo supplement (microcrystalline cellulose). Both groups received a container with the product and a dosing measure (5 g). The intervention was developed for 12 weeks. Blood samples and stools were taken at the beginning and end of the intervention.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beta-Glucan (BETA) (Experimental): experimental group, received a supplement of oats beta-glucan (5 g) for 12 weeks.
  Interventions: Dietary Supplement: Oat Beta-glucan as a Supplement in Type 2 Diabetics
- Control (CN) (Placebo Comparator): placebo group, received a supplement of cellulose microcrystalline (5g) for 12 weeks.
  Interventions: Dietary Supplement: Oat Beta-glucan as a Supplement in Type 2 Diabetics

INTERVENTIONS:
Dietary Supplement: Oat Beta-glucan as a Supplement in Type 2 Diabetics — 44 subjects were randomized into two groups, placebo (PL) and β-glucan (BG). Each person received a package with a supplement sufficient for 12 weeks, adding 5 g of supplement to breakfast, which could contain beta-glucan or not. Blood and stool samples were requested at the beginning and at the end of the intervention.

SUMMARY:
Objective: To evaluate the effect of oat β-glucans on the satiety perception, metabolic control and intestinal microbiota of type 2 diabetics from Talca, Chile. Methodology: Clinical trial, controlled, randomized, double blind and parallel design. The recruited (40 subjects) were randomized into two groups, placebo (PL) and ß-glucan (BG). 5 gr of oat ß-glucan or placebo were delivered for 12 weeks to be added in breakfast. Blood and stool samples were requested at the beginning and at the end of the intervention. The investigators quantify: HbA1c in whole blood, fasting blood glucose, basal insulin, C-peptide, tumor necrosis factor alpha (TNF-a), interleukin (IL) 6, IL-8, IL-10, IL1β, cortisol, ghrelin, glucagon-like peptide type 1 (GLP -1), YY peptide (PYY), Resistin, Leptin and serum Lipid Profile. The subjective perception of hunger / satiety were established through an analogous visual survey. Calorie intake was determined by 24-hour recall survey. Were analyzed the phylum: Firmicutes, Bacteroidetes and Verrucomicrobia, and the populations of Bifidobacteria spp, Lactobacillus spp, butyrate producing bacteria, Akkermansia Muciniphila and total bacteria of fecal microbiota, using quantitative polymerase chain reaction (qPCR) with specific primers. All participants were instructed not to make changes in their usual eating habits, physical activity and pharmacological treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes mellitus
* Use of oral hypoglycemic agents (Metformin)
* 30 to 45 years
* More than one year and less than 10 diabetes
* no major chronic complications
* Hb A1c between 7 to 9%
* BMI between 30-35 Kg / mt2.

Exclusion Criteria:

* Pregnant women
* Acute and / or chronic intestinal pathologies (malabsorption syndrome, celiac disease, chronic inflammatory bowel diseases, among others.),
* Drugs that interfere with the microbiota (antibiotics, anti-inflammatories, laxatives, prokinetics),
* Organic insufficiencies (cardiac, hepatic, renal, respiratory), or with immunodeficiencies (HIV, chemotherapy, radiotherapy, transplanted).
* Presence of smoking habit.
* Regular probiotic or prebiotic intake (more than 2 months)
* Dipeptidyl peptidase 4 inhibitors (DPP4) and α-amylase inhibitor drugs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2019-01-18 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks
  Concentration of Glycated Hemoglobin A

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Estudios en Alimentación y Nutrición, Talca, Maule Region, Chile

REFERENCES:
- [Background] Francelino Andrade E, Vieira Lobato R, Vasques Araujo T, Gilberto Zangeronimo M, Vicente Sousa R, Jose Pereira L. Effect of beta-glucans in the control of blood glucose levels of diabetic patients: a systematic review. Nutr Hosp. 2014 Jan 1;31(1):170-7. doi: 10.3305/nh.2015.31.1.7597. PMID 25561108
- [Background] Abbasi NN, Purslow PP, Tosh SM, Bakovic M. Oat beta-glucan depresses SGLT1- and GLUT2-mediated glucose transport in intestinal epithelial cells (IEC-6). Nutr Res. 2016 Jun;36(6):541-52. doi: 10.1016/j.nutres.2016.02.004. Epub 2016 Feb 18. PMID 27188900
- [Background] Beck EJ, Tosh SM, Batterham MJ, Tapsell LC, Huang XF. Oat beta-glucan increases postprandial cholecystokinin levels, decreases insulin response and extends subjective satiety in overweight subjects. Mol Nutr Food Res. 2009 Oct;53(10):1343-51. doi: 10.1002/mnfr.200800343. PMID 19753601
- [Background] Dong J, Cai F, Shen R, Liu Y. Hypoglycaemic effects and inhibitory effect on intestinal disaccharidases of oat beta-glucan in streptozotocin-induced diabetic mice. Food Chem. 2011 Dec 1;129(3):1066-71. doi: 10.1016/j.foodchem.2011.05.076. Epub 2011 May 25. PMID 25212338
- [Background] Pentikainen S, Karhunen L, Flander L, Katina K, Meynier A, Aymard P, Vinoy S, Poutanen K. Enrichment of biscuits and juice with oat beta-glucan enhances postprandial satiety. Appetite. 2014 Apr;75:150-6. doi: 10.1016/j.appet.2014.01.002. Epub 2014 Jan 14. PMID 24434584
- [Background] Shen XL, Zhao T, Zhou Y, Shi X, Zou Y, Zhao G. Effect of Oat beta-Glucan Intake on Glycaemic Control and Insulin Sensitivity of Diabetic Patients: A Meta-Analysis of Randomized Controlled Trials. Nutrients. 2016 Jan 13;8(1):39. doi: 10.3390/nu8010039. PMID 26771637